CLINICAL TRIAL: NCT04487990
Title: CoV-Hep Study: Randomized and Paired Clinical Trial Comparing Regional Anticoagulation Modalities in Continuous Venous Venous Hemodialysis in Patients With COVID-19
Brief Title: CoV-Hep Study: Regional Anticoagulation Modalities in Continuous Venous Venous Hemodialysis in Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1252-0194; 33351120.0.0000.0068 (Other: CAAE / CONEP / CEP)
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Acute Kidney Injury; Covid19
Keywords: acute kidney injury; continuous venovenous hemodialysis; anticoagulation; heparin; citrate; covid-19
MeSH Terms: conditions — Acute Kidney Injury; COVID-19 | interventions — Heparin

STUDY DESIGN:
Intervention Model Description: Clinical trial of treatment, randomized-controlled, parallel, open, with two arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Patients on continuous hemodialysis (blood flow 150 ml / min, dose of 30 ml / kg / h) receiving anticoagulation with sodium citrate at 4 mmol / l.
- Intervention group (Experimental): Patients on continuous hemodialysis (blood flow 150 ml / min, dose of 30 ml / kg / h) receiving anticoagulation with sodium citrate at 4 mmol / l associated with unfractionated heparin at 10U / Kg / h.
  Interventions: Drug: unfractionated Heparin

INTERVENTIONS:
Drug: unfractionated Heparin — Addition of unfractioned heparin to CVVHD system already running under citrate regional anticoagulation.
  Other Names: No associated drug
  Arms: Intervention group

SUMMARY:
Since the emergence of the new strain of betacoronavirus (SARS-CoV-2) and its important clinical repercussions, it has been described that patients with its associated pneumonia (COVID-19) have high rates of thrombotic events, including reduction in the dialyzers patency when undergoing renal replacement therapy. Several strategies for preventing the early loss of dialysers are described, and regional anticoagulation based on citrate is the preferred modality for preventing this complication. On the other hand, in patients with SARS-CoV-2 there are already descriptions of endothelial inflammation and activation of the coagulation cascade, including studies demonstrating the benefit of heparinization of these patients. Thus, this study aims to compare two different anticoagulation strategies in patients infected with COVID-19 with continued venovenous hemodialysis (CVVHD). From the indication of CVVHD, patients will be screened according to eligibility criteria and, if they fit these parameters, they will be randomized into two groups: Group A - Standard regional anticoagulation based on Citrate associated with infusion of low doses of unfractionated heparin 10ui/kg/hour and Group B - Standard regional anticoagulation based on Citrate only. Patients will be randomized in blocks and followed for 72 hours. The primary endpoint is dialyzer patency at the end of 72 hours of clinical follow-up. Secondary objectives will be mortality, bleeding rate, drop in hematimetric indices, urea sieving, filter time in hours, down time of therapy, system and dialyser pressures (PBE and PTM). All patients will undergo a standard procedure with a prescribed dose of 30mL/Kg/H, blood flow of 150mL/minute and polysulfone dialyzer.

DETAILED DESCRIPTION:
After randomization, patients will be allocated to one of two groups:

Control group (n = 45): patients on continuous hemodialysis (blood flow 150 ml / min, dose of 30 ml / kg / h) receiving anticoagulation with sodium citrate at 4 mmol / l. The dialysis system pressures, dialyzer patency and duration and bleeding rate will be assessed for 72 hours;

Intervention group (n = 45): patients on continuous hemodialysis (blood flow 150 ml / min, dose of 30 ml / kg / h) receiving anticoagulation with sodium citrate at 4 mmol / l associated with unfractionated heparin at 10U / Kg / h. The dialysis system pressures, dialyzer patency and duration and bleeding rate will be assessed for 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or probable SARS-CoV-2 infection;
* Presence of acute kidney injury with indication and agreement between ICU and nephrology teams for the introduction of renal continuous venous venous hemodialysis.

Exclusion Criteria:

* Hypersensitivity to any of the substances used in the study (Citric acid dextrosol 2.2% and unfractionated heparin);
* Previous diagnosis of coagulopathy or thrombophilia;
* Contraindication to the use of unfractionated heparin by the assistant team;
* Risk of citrate poisoning - (Lactate> 30mg / dL, RNI> 2.5, Total bilirubin> 15mg / dL);
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-03 (Actual)

PRIMARY OUTCOMES:
Clotted dialyzers | Day 3 of dialysis
  The percentage of clotted dialyzers within 72 hours in each of the studied groups.

SECONDARY OUTCOMES:
Time-free of clotting | Day 3 of dialysis
  Number of hours until a dialyzer clots in the first 72 hours of dialysis
Number of dialyzers used | Day 3 of dialysis
  The amount of dialyzers used in the first 72 hours of hemodialysis
Pressure variation | Day 3 of dialysis
  Variation in dialysis system and vascular access pressures in the first 72 h of dialysis
Urea sieving | Day 3 of dialysis
  Variation in urea sieving between the first, second and third days of dialysis
Downtime of dialysis | Day 3 of dialysis
  Time of dialysis stop due to clotting in the first 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Lins, MD, Principal Investigator — University of São Paulo General Hospital; Camila Rodrigues, MD, PhD, Principal Investigator — University of São Paulo General Hospital
Locations (1):
- University of São Paulo General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Lins PRG, de Albuquerque CCC, Assis CF, Rodrigues BCD, E Siqueira Campos BP, de Oliveira Valle E, Cabrera CPS, de Oliveira Gois J, Segura GC, Strufaldi FL, Mainardes LC, Ribeiro RG, Via Reque Cortes DDP, Lutf LG, de Oliveira MFA, Sales GTM, Smolentzov I, Reichert BV, Andrade L, Seabra VF, Rodrigues CE. Cov-hep study: heparin in standard anticoagulation based on citrate for continuous veno-venous hemodialysis in patients with COVID-19: a structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Nov 11;21(1):920. doi: 10.1186/s13063-020-04814-0. PMID 33176886